CLINICAL TRIAL: NCT07203404
Title: A Clinical Study of the Safety, Efficacy, and Cell Pharmacokinetics of Anti-CD19/BCMA Universal CAR-T Cell Therapy RD06-05 in Patients With Autoimmune Diseases.
Brief Title: A Study of Anti-CD19/BCMA Universal CAR-T Cell Therapy RD06-05 in Patients With Autoimmune Diseases.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD06-05
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: SLE; LN; ANCA Associated Vasculitis; ANCA-Associated Glomerulonephritis; Anti-GBM Disease; MN; SSc; IIM
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Anti-Glomerular Basement Membrane Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD06-05 (Experimental)
  Interventions: Drug: RD06-05 CART Cell Injection

INTERVENTIONS:
Drug: RD06-05 CART Cell Injection — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide

SUMMARY:
An Exploratory, Single-Arm, Open-Label, Dose-Escalation Study of the Safety, Tolerability, PK, PD, and Efficacy of Anti-CD19/BCMA Universal CAR-T Therapy RD06-05 in Autoimmune Diseases (including SLE/LN, AAV/AAGN, Anti-GBM, MN, SSc, and IIM).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Aged ≥18 years and ≤75 years.
3. Adequate organ function defined as:

   1. Bone marrow function: Defined as absolute neutrophil count (ANC) ≥1500/μL, absolute lymphocyte count (ALC) ≥100/μL, hemoglobin (Hb) ≥80 g/L, and platelet count (PLT) ≥50,000/μL. Transfusions and growth factors must not have been used within 7 days prior to screening to meet these criteria.
   2. Liver function: Defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN), and total bilirubin <1.5 × ULN (or <3.0 × ULN for subjects with Gilbert's syndrome).
   3. Coagulation function: Defined as international normalized ratio (INR) or partial thromboplastin time (PTT) ≤1.5 × ULN.
   4. Pulmonary function: Defined as dyspnea ≤ Grade 1 per CTCAE and oxygen saturation (SpO₂) ≥92% on room air (by pulse oximetry).
4. Female subjects of childbearing potential must have a negative serum or urine pregnancy test. Females who are surgically sterile or postmenopausal for at least 2 years are considered not of childbearing potential.
5. From the time of signing the informed consent form until 6 months after the completion of RD06-05 infusion, female subjects of childbearing potential and male subjects with partners of childbearing potential must use highly effective methods of contraception.

Inclusion Criteria for Subjects with Anti-GBM Disease:

Diagnosis of anti-GBM disease according to the 2012 Chapel Hill Consensus Conference definitions, meeting both of the following criteria:

1. Positive for anti-GBM antibody (based on historical or screening test results);
2. Evidence of renal involvement at screening, defined as:

   1. Presence of active, pathologically confirmed anti-GBM disease (renal biopsy must have been performed within 1 year prior to the screening visit or during the screening period); and
   2. Accompanied by proteinuria and hematuria.

Inclusion Criteria for Subjects with SLE/LN:

1. Diagnosis of SLE according to the 2019 European Alliance of Associations for Rheumatology (EULAR)/American College of Rheumatology (ACR) classification criteria or the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria.
2. Positive for antinuclear antibody (ANA), and/or anti-double-stranded DNA (anti-dsDNA) antibody, and/or anti-Smith (anti-Sm) antibody at screening.
3. SLEDAI-2K score > 6 points at screening.

Inclusion Criteria for Subjects with AAV/AAGN:

1. Diagnosis of microscopic polyangiitis (MPA) or granulomatosis with polyangiitis (GPA) according to the 2022 ACR/EULAR classification criteria for ANCA-associated vasculitis.
2. Positive for anti-myeloperoxidase (MPO-ANCA) antibody or anti-proteinase 3 (PR3-ANCA) antibody at screening or based on historical testing.
3. For AAV without renal involvement: A Birmingham Vasculitis Activity Score (BVAS) version 3 score of ≥3 at screening, indicating active vasculitis.

Inclusion Criteria for Subjects with MN:

1. Diagnosis of primary (idiopathic) membranous nephropathy confirmed by renal biopsy pathology (the renal biopsy must have been performed within 2 years prior to screening or during the screening period).
2. Meeting the criteria for high-risk or relapsed/refractory membranous nephropathy:

High-risk patients, defined as meeting any of the following criteria:

1. Normal eGFR with urine protein >3.5g/24h, a reduction of <50% in urine protein after 6 months of ACEI/ARB treatment, and serum albumin <25 g/L or anti-PLA2R antibody >50 RU/mL;
2. eGFR <60 mL/min/1.73m² and/or urine protein >8g/24h for more than 6 months.

Refractory/Relapsed patients:

Refractory patients are defined as those resistant to prior immunosuppressive therapy (persistent urine protein ≥3.5g/24h with a <50% reduction from baseline).

Relapsed patients are defined as those who achieved complete or partial remission with prior immunosuppressive therapy but subsequently developed recurrent urine protein ≥3.5g/24h.

Inclusion Criteria for Subjects with SSC:

1. Diagnosis of systemic sclerosis (SSc) according to the 2013 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology (EULAR) classification criteria.
2. Diagnosis of diffuse cutaneous SSc at screening.

Inclusion Criteria for Subjects with IIM:

1.Diagnosis of idiopathic inflammatory myopathy (IIM) according to the 2017 ACR/EULAR classification criteria (including probable or definite diagnosis, corresponding to a probability score of ≥55%). The subtypes include dermatomyositis (DM), anti-synthetase syndrome (ASS), and immune-mediated necrotizing myopathy (IMNM).

Exclusion Criteria:

1. Subjects with SLE/LN:

   1. Severe active central nervous system (CNS) lupus, including psychosis, seizures, lupus headache, or other signs/symptoms associated with neuropsychiatric lupus, as assessed by a qualified specialist during screening.
   2. Drug-induced or secondary lupus.
2. Subjects with AAV/AAGN:

   1. Drug-induced or secondary AAV/AAGN.
   2. Presence of alveolar hemorrhage requiring invasive ventilatory support at screening.
3. Subjects with Anti-GBM Disease:

   1. Anuria for more than 7 days.
   2. Dialysis dependence for more than 30 days.
   3. Ongoing moderate or severe pulmonary hemorrhage (or cessation within the past two weeks) defined as pulmonary hemorrhage requiring assisted ventilation, supplemental oxygen, or blood transfusion.
   4. Symptomatic congestive heart failure (NYHA Class 2-4) requiring prescription medication or clinically significant cardiogenic peripheral edema.
4. Subjects with MN:

   Secondary membranous nephropathy.
5. Subjects with IIM:

   Presence of severe rhabdomyolysis or CK level ≥120 × ULN at screening.
6. Subjects with SSc:

   1. History of scleroderma renal crisis within 1 year prior to screening.
   2. History of cardiac tamponade within 6 months prior to screening.
   3. Active infection of digital ulcers within 3 months prior to screening.
   4. Presence of digital gangrene at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-07-23 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (TEAEs), serious adverse events (SAEs), and adverse events of particular concern (AESI) during treatment | 2 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Bioheng Study site, Shanghai, China